CLINICAL TRIAL: NCT07077915
Title: Osseodensification vs Conventional Drilling for Immediate Dental Implant Placement: A Randomized Controlled Clinical and Radiographic Study
Brief Title: Osseodensification vs Conventional Drilling for Immediate Dental Implant Placement
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamad Ali Itani (Other)
Collaborators: Beirut Arab University (Other)
Responsible Party: Sponsor-Investigator, Mohamad Ali Itani, Master of Science candidate in Periodontics, Beirut Arab University
Organization: Beirut Arab University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-H-0162-D-M-0696
Record Dates: First submitted 2025-07-12; First posted 2025-07-22 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Immediate Dental Implant Placement; Conventional Drilling Technique; Osseodensification Drilling Technique
Keywords: immediate dental implant; immediate dental implant with bone graft; osseodensification; conventional drilling; densah burs

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Osseodensification burs (Experimental)
  Interventions: Other: Osseodensification burs
- Conventional Burs (Active Comparator)
  Interventions: Other: Conventional burs

INTERVENTIONS:
Other: Osseodensification burs — Densah burs are osseodensification burs used to condense bone and prepare dental implant site, unlike conventional technique which cuts and removes the bone
  Arms: Osseodensification burs
Other: Conventional burs — Preparation of dental implant site by the Conventional technique using Conventional burs that are subtractive
  Arms: Conventional Burs

SUMMARY:
Aim of the study is to analyze and compare the characteristic differences occurring in the surrounding bone in an immediate implant placed by osseodensification to immediate implants placed with the conventional technique

DETAILED DESCRIPTION:
A bifurcation inter-radicular bone of 2 mm or more in a none restorable lower molar will be needed in order to successfully be able to drill the bone with conventional or Osseo densification burs, followed by placing the implant at this site. A xenograft bone material will be used to fill the extraction socket and a customized temporary abutment using flowable composite and a silicone mold will be fabricated and placed over it after polishing it.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age 25 to 45 years old
2. Systemically and periodontally healthy individuals.
3. Non-smokers or light smokers (Less than 5 cigarettes a day) (Schane 2010).
4. Good oral hygiene.
5. Healthy remaining dentition.
6. Adequate quality and quantity of bone
7. Interradicular septum ≥ 2 mm (Bleyan, 2022).
8. Mandibular non-restorable molars.
9. Type A or B socket (Smith and Tarnow, 2013).

Exclusion Criteria:

1. Acute inflammation or infection in the implant region.
2. Patients with mental disorders who could not cooperate with treatment or communicate normally.
3. Patients who have severe systemic disorders (Uncontrolled Diabetes, Uncontrolled Hypertension, End stage kidney or liver diseases and Severe Heart diseases) .
4. Poor oral hygiene.
5. Active periodontal disease.
6. Uncooperative patients, not willing to adhere to post-surgical instructions and follow up visits.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12-23 (Estimated); Study Completion 2025-12-23 (Estimated)

PRIMARY OUTCOMES:
Interradicular bone width | Intraoperative (at time of surgery)
  The width of the interradicular bone in the interradicular septum will be measured immediately before and after drilling is performed during surgery. Measurements will be taken using a UNC-15 periodontal probe and recorded in millimeters (mm).
Dental implant stability | up to 4 months after dental implant placement
  Implant stability will be assessed using the Osstell device, which uses resonance frequency analysis to calculate an Implant Stability Quotient (ISQ). ISQ values range from 1 to 100, with higher values indicating greater implant stability.

SECONDARY OUTCOMES:
Marginal Bone Level | up to 7 months after the implantation
  Bone levels will be estimated on the labial, palatal, distal, and mesial surfaces of each implant using cone-beam computed tomography (CBCT). Measurements will be taken from a fixed reference point at the implant shoulder to the bone crest. All measurements will be recorded in millimeters (mm).
Bone density | up to 7 months after dental implant placement
  Bone density will be measured in four regions around each dental implant: buccal, lingual, apical, and crestal. The mean grayscale value for each implant will be calculated based on these four areas. Bone density values will be obtained from cone-beam computed tomography (CBCT) and expressed in grayscale units.

CONTACTS AND LOCATIONS:
Overall Officials: Nayer Aboelsaad, Phd, Study Chair — Beirut Arab Univeristy; Rania Abdelaziz, Phd, Study Director — Beirut Arab University; Hani Arakji, Phd, Study Director — Beirut Arab University
Locations (1):
- Beirut Arab University, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] https://omx.journals.ekb.eg/article_140845_40c7deeba68c3279a9d3dffaed37c3fd.pdf
- See also: This article includes information about the success and stability achieved by using osseodensification technique — https://jcdr.net/article_fulltext.asp?id=11749
- See also: This article includes information regarding stability of dental implants in narrow ridges when using conventional burs and osseodensifications burs — https://pdfs.semanticscholar.org/108e/c798b9f6cb0eb4a2888840f962adf0ffdc89.pdf
- See also: This study includes information about marginal bone level and dental implant stability in conventional vs osseodensification techniques — https://journals.lww.com/jips/fulltext/2020/20010/to_compare_the_stability_and_crestal_bone_loss_of.7.aspx